CLINICAL TRIAL: NCT03664609
Title: Deep Brain Stimulation (DBS) Retrospective Outcomes Study
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A4170
Record Dates: First submitted 2018-08-31; First posted 2018-09-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Parkinson Disease; Essential Tremor; Dystonia
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Parkinson's Disease: Subjects with Parkinson's disease, implanted with a Boston Scientific Deep Brain Stimulation System
  Interventions: Device: Deep Brain Stimulation
- Essential Tremor: Subjects with Essential Tremor, implanted with a Boston Scientific Deep Brain Stimulation System
  Interventions: Device: Deep Brain Stimulation
- Dystonia: Subjects with dystonia, implanted with a Boston Scientific Deep Brain Stimulation System
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation in patients with Parkinson Disease, Dystonia and Essential Tremor.

SUMMARY:
The primary objective of this study is to characterize real-world clinical outcomes of Deep Brain Stimulation (DBS) using retrospective review of de-identified patient records.

DETAILED DESCRIPTION:
The purpose of this study is to characterize

1. real-world clinical outcomes of Deep Brain Stimulation (DBS) using retrospective review of de-identified patient records.

ELIGIBILITY:
Inclusion Criteria:

* Must be previously treated with or eligible for implantation with a deep brain stimulation system

Exclusion Criteria:

* No Exclusion Criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects' chart data will be drawn from the Investigator's standard patient pool treated at his/her practice.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Unified Parkinson's Disease Rating Scale (UPDRS III) at up to 5 years post implant compared to baseline | 5 yrs. post implant
  Improvement in disease symptoms as assessed by Unified Parkinson's Disease Rating Scale (UPDRS III) at up to 5 years post implant compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Neuromodulation Corporation
Locations (19):
- United States (9):
  - St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - University of Miami Hospital, Miami, Florida
  - University of South Florida, Tampa, Florida
  - St. Luke's Regional Medical Center, Boise, Idaho
  - Albany Medical Center, Albany, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Swedish Neuroscience Institute, Seattle, Washington
- Belgium (2):
  - AZ St. Lucas, Ghent
  - AZ Delta, Roeselare
- Hopital Fondation Adolphe de Rothschild, Paris, France
- Germany (5):
  - Uniklinik Köln, Cologne
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - Uniklinikum Jena, Jena
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - Universitaetsklinikum Wuerzburg, Würzburg
- Fondazione Istituto Neurologico Casimiro Mondino, Pavia, Italy
- Hospital Virgen Del Rocio, Seville, Spain

IPD SHARING:
Plan to Share IPD: No